CLINICAL TRIAL: NCT06110260
Title: Pharmacokinetic Effect of AstraGin on Whey Protein Absorption and Muscle Function in Healthy Subjects: A Randomized, Double-blind, Crossover Trial.
Brief Title: Pharmacokinetic Effect of AstraGin on Whey Protein Absorption and Muscle Function in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: CS1-23151
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pharmacokinetic Effect of AstraGin on Whey Protein Absorption and Muscle Function in Healthy Subjects
Keywords: BCAA; Ginseng and Astragalus Saponin Extract; Whey Protein; Pharmacokinetics
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AstraGin (Experimental): The 1st round: Before each study day, all subjects took a 50 mg AstraGin capsule at 9 p.m. and began fasting for 12 hours, except for a small amount of water the night before the experiment. On each study day, all subjects collected their first blood sample at 9 a.m. from the median cubital vein using the indwelling catheter method. After the first blood collection, all subjects took 50 mg AstraGin and 35 g of whey protein with 250 mL water.
  Additional blood samples were collected at 0, 15, 30, 45, 60, 90, 120, 150, and 180 min to analyze the plasma concentration of amino acids.
  The washout period is seven days, during which the subjects maintain a stable lifestyle and dietary habits.
  The 2nd round: All subjects take a 50 mg AstraGin capsule and conduct the procedure (same as the 1st round)
  Interventions: Dietary Supplement: AstraGin (Ginseng and Astragalus Saponin Extract)
- Placebo (Placebo Comparator): The 1st round: Before each study day, all subjects took a 50 mg placebo (maltodextrin) capsule at 9 p.m. and began fasting for 12 hours, except for a small amount of water the night before the experiment. On each study day, all subjects collected their first blood sample at 9 a.m. from the median cubital vein using the indwelling catheter method. After the first blood collection, all subjects took 50 mg placebo and 35 g of whey protein with 250 mL water.
  Additional blood samples were collected at 0, 15, 30, 45, 60, 90, 120, 150, and 180 min to analyze the plasma concentration of amino acids.
  The washout period is seven days, during which the subjects maintain a stable lifestyle and dietary habits.
  The 2nd round: All subjects take a 50 mg Placebo capsule and conduct the procedure (same as the 1st round)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AstraGin (Ginseng and Astragalus Saponin Extract) — In this study, we are investigating the effects of AstraGin on healthy adults. The testing sample is orally administrated to subjects with 35g whey protein + AstraGin. After intervention, a 180-min kinetics study of plasma amino acids was conducted.
  Arms: AstraGin
Dietary Supplement: Placebo — In this study, we are investigating the effects of AstraGin on healthy adults. The testing sample is orally administrated to subjects with 35g whey protein + Placebo. After intervention, a 180-min kinetics study of plasma amino acids was conducted.
  Arms: Placebo

SUMMARY:
This study gave healthy people supplements with ginseng and astragalus saponin extracts (AstraGin), combined with whey protein, to explore whether it can promote amino acid absorption and thereby enhance protein nutritional status and muscle function.

This trial is a randomized, double-blind, crossover trial, and the research subjects are adult healthy subjects.

DETAILED DESCRIPTION:
A randomized-double blind, crossover human trial. 30 healthy adults, subdivided into two groups, are randomized into treatments and placebo groups to ensure equally balanced randomization and comparability, considering factors including age, sex, and diet.

(2) The 1st round: Before each study day, all subjects took a 50 mg AstraGin/placebo (maltodextrin) capsule at 9 p.m. and began fasting for 12 hours, except for a small amount of water the night before the experiment. On each study day, all subjects collected their first blood sample at 9 a.m. from the median cubital vein using the indwelling catheter method. After the first blood collection, all subjects took 50 mg AstraGin/placebo and 35 g of whey protein with 250 mL water.

(3) Additional blood samples were collected at 0, 15, 30, 45, 60, 90, 120, 150, and 180 min to analyze the plasma concentration of amino acids.

(5) The washout period is seven days, during which the subjects maintain a stable lifestyle and dietary habits. The 2nd round: All subjects take a 50 mg Placebo/AstraGin capsule and conduct the procedure (same as the 1st round)

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults and aged 20-65 years.
* Subject has provided written informed consent to participate in the study.
* The subject is willing and able to comply with the study.

Exclusion Criteria:

* The subject is participating in another clinical trial thirty days prior to enrollment.
* Subject allergy to milk proteins
* Subject has diabetes, obesity, hypertension, cardiovascular disease, liver or kidney disease, current infections, and smoking were exclusion criteria.
* Subject has any medical condition or uses any medication, nutritional product, amino acids supplement, or program which might interfere with the conduct of the study or place the subject at risk.
* Subjects lost to follow-up, non-compliance, and concomitant medication.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
The AUC of BCAA in human plasma | 3 hr
  Pharmacokinetic ( 0, 15, 30, 45, 60, 90, 120, 150, and 180 minutes)

SECONDARY OUTCOMES:
Plasma TAC Test | 4weeks、12weeks
Grip Strength | 4weeks、12weeks
  Handgrip strength is assessed using a hand dynamometer to evaluate muscle strength
Muscle Mass-DXA | 4weeks、12weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Shan Medical University, Taichung, Taiwan